CLINICAL TRIAL: NCT07131930
Title: The Relationship Between Caregiver Burden, Resilience Level and Sleep Quality in Individuals Providing Care for Bedridden Patients
Brief Title: A Study on the Relationship Between Caregiver Burden, Resilience, and Sleep Quality in Individuals Providing Care for Bedridden Patients
Acronym: Caregiver
Status: Completed | Type: Observational
Sponsor: UĞUR UZUN (Other)
Collaborators: Tepecik Training and Research Hospital (Other)
Responsible Party: Sponsor-Investigator, UĞUR UZUN, Specialist in Anesthesiology and Reanimation, Tepecik Training and Research Hospital
Organization: Tepecik Training and Research Hospital (Other)
Other Study IDs: 2023/09-20; 2023/09-20 (Registry Identifier: Ethics Committee Approval Number: 2023/09-20-Tepecik Training and Research Hospital)
Record Dates: First submitted 2025-08-04; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: Caregiver Burden
Keywords: Caregiver Burden; Resilience; Sleep Quality; Palliative Care
MeSH Terms: conditions — Caregiver Burden; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Caregiver Burden, Psychological Resilience, Sleep Quality — Informal caregivers who provide daily care for bedridden patients are evaluated in this study. The exposure involves physical, emotional, and financial caregiving responsibilities such as assistance with feeding, mobility, and emotional support. The impact of caregiving on sleep quality and psychological resilience is assessed using validated questionnaires (Zarit Burden Interview, Pittsburgh Sleep Quality Index, Resilience Scale).

SUMMARY:
This observational study aims to examine the relationship between caregiver burden, psychological resilience, and sleep quality in individuals providing care for bedridden patients, particularly in the context of palliative care. In many cases, the care of bedridden patients in hospitals and at home is undertaken by family members. The caregiving process can be physically, emotionally, and financially demanding. Caregivers often face challenges such as irregular eating habits, chronic fatigue, body pain, difficulty concentrating, restlessness, insomnia, and even increased use of alcohol or medication. These burdens can also negatively impact their social relationships, work performance, and financial stability.

As caregiver burden increases, caregivers are more likely to experience sleep disorders, anxiety, depression, stress, and burnout. These issues not only affect the caregiver's quality of life but also reduce the quality of care provided to the patient. It is therefore crucial to assess the psychosocial needs of caregivers and to understand the factors that influence their ability to cope with caregiving demands.

Psychological resilience-defined as the ability to adapt to stress and recover from adversity-is believed to play a key role in coping with caregiver stress, though its relationship with caregiver burden remains unclear. This study will evaluate caregiver burden, sleep quality, and psychological resilience using validated questionnaires. Participants will be caregivers of patients currently hospitalized in our palliative care unit. After obtaining ethical approval, individuals who consent to participate will complete the questionnaires. The results will help inform future support strategies aimed at improving caregiver well-being and patient care quality.

DETAILED DESCRIPTION:
This observational study is conducted to evaluate the relationship between caregiver burden, psychological resilience, and sleep quality among individuals providing care for bedridden patients in a hospital-based palliative care unit.

The study population will consist of caregivers (aged 18 and older) of patients hospitalized in the palliative care unit. After obtaining ethics committee approval, voluntary participants who provide informed consent will be asked to complete a series of validated self-report questionnaires, including:

* Zarit Burden Interview (ZBI) to assess caregiver burden
* Pittsburgh Sleep Quality Index (PSQI) to measure sleep quality
* Resilience Scale to assess psychological resilience The sample size was estimated based on similar studies in the literature, aiming for a minimum of 100 participants to achieve sufficient statistical power. Statistical analysis will be performed using SPSS software (v27). Descriptive statistics, correlation analysis, and multiple linear regression models will be used to examine the relationships among caregiver burden, sleep quality, and resilience. A p-value of <0.05 will be considered statistically significant.

The data will be collected through face-to-face interviews or self-administered paper questionnaires. Participants' sociodemographic characteristics will also be recorded. The study does not involve any interventions or experimental procedures.

Findings from this study may contribute to the development of targeted psychosocial interventions to support caregivers of functionally dependent patients and improve the overall quality of care.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older
* Informal caregivers (family members or close contacts) providing daily care for bedridden patients hospitalized in the palliative care unit
* Ability to provide informed consent
* Willingness to voluntarily participate in the study

Exclusion Criteria:

* Individuals under the age of 18
* Individuals with cognitive impairments that prevent them from completing the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Informal caregivers of bedridden patients who are currently hospitalized in the palliative care unit of a tertiary care hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Correlation between Zarit Burden Interview (ZBI, 19-item scale) and Adult Resilience Scale (ARS, 33-item scale) | at enrollment

SECONDARY OUTCOMES:
Correlation between Zarit Burden Interview (ZBI, 19-item scale) and Pittsburgh Sleep Quality Index (PSQI, 19-item scale) | At enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Tepecik Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No